CLINICAL TRIAL: NCT00113230
Title: Phase II Trial Of Neoadjuvant Concurrent Capecitabine, RHUMAB VEGF (Avastin) And Radiotherapy In Patients Presenting With Locally Advanced Rectal Cancer
Brief Title: Neoadjuvant Chemoradiation With RHUMAB VEGF (Avastin) for Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0832
Record Dates: First submitted 2005-06-06; First posted 2005-06-07 (Estimated); Results first posted 2009-11-13 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-07

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Bevacizumab; RHUMAB VEGF; Avastin; Capecitabine; Neoadjuvant Concurrent Capecitabine; Xeloda; Radiation; Radiotherapy; Radiation Therapy; XRT
MeSH Terms: conditions — Rectal Neoplasms | interventions — Bevacizumab; Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Avastin (Experimental): Capecitabine, Avastin (RHUMAB VEGF/Bevacizumab) And Radiotherapy
  Interventions: Drug: Avastin (Bevacizumab, RHUMAB VEGF); Drug: Capecitabine; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Avastin (Bevacizumab, RHUMAB VEGF) — Starting Dose 5 mg/kg intravenously on day one of radiotherapy, given every 2 weeks +/- 2 days for a total of 3 doses.
  Other Names: RHUMAB VEGF; Avastin; Bevacizumab
Drug: Capecitabine — 900 mg/m^2 by mouth twice a day during days of radiation for all five weeks of therapy.
  Other Names: Xeloda
Radiation: Radiation Therapy — 45 Gy in 25 fractions to the pelvis followed by 5.4 Gy as a boost dose to the primary tumor with margin, for a total dose of 50.4 Gy over 28 treatment days.
  Other Names: XRT; Radiotherapy

SUMMARY:
Preoperative chemoradiation leads to increased pelvic control and overall survival, but both distant and local disease control remain problematic in locally advanced rectal cancer patients. Enhancing the effect of chemotherapy and radiotherapy can increase tumor response as well as distant disease control. Patients who have complete response to therapy have increased sphincter preservation, and can possibly have more limited surgery (full thickness local excision). When combined with standard chemotherapy, bevacizumab [RHUMAB VEGF, Avastin] has been shown to improve response and median survival in patients with metastatic colorectal cancer in a recent randomized trial, has led to increased activity in preclinical studies with radiotherapy, and has been found to be very well tolerated with chemoradiation in a phase I trial conducted at the M.D. Anderson Cancer Center (MDACC) in patients with locally advanced pancreatic cancer. The hypothesis is that the addition of bevacizumab to standard chemoradiation will safely lead to increased tumor response in patients with locally advanced rectal cancer.

DETAILED DESCRIPTION:
Avastin [RHUMAB VEGF, Bevacizumab] is a drug that has damaging effects on blood vessel growth in tumors.

Before treatment starts, you will have a complete physical exam. About 2 tablespoons of blood will be drawn for routine tests and a urine test will be performed. Chest x-rays and CT scans of the abdomen and pelvis will be done. Women who are able to have children must have a negative blood pregnancy test.

You will receive radiation therapy once a day for 5 days in a row (Monday-Friday) for 5 weeks and three days (a total of 28 treatments). You will take the chemotherapy drug capecitabine by mouth twice a day on each of the days that you receive radiation therapy. These pills will not be taken on Saturday and Sunday. You must not take cimetidine, and must be off of coumadin for at least one week and sorivudine and brivudine for at least four weeks before starting capecitabine and while taking capecitabine.

You will receive the drug Avastin by vein once every 2 weeks for six weeks (a total of three doses). The infusion will at first last 90 minutes. If there are no allergic reactions, fevers or chills, it will be shortened to 60 minutes and then 30 minutes for later infusions.

During the study, you will have physical exams, including weekly blood tests (about 2 teaspoons). The possible development of side effects will be closely monitored.

All participants will have surgical removal of the rectal tumor 6-8 weeks after the completion of treatment as they would for the standard of care for their disease. No patients will have surgery before 6 weeks.

After participation in this study is over, you will have follow-up evaluation as needed for standard of care.

THIS IS AN INVESTIGATIONAL STUDY. Capecitabine is approved by the FDA, but Avastin has not yet been evaluated for approval.

About 50 patients will take part in the study. All will be enrolled at the M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG status of 0 or 1.
2. Patients must be greater than or equal to 18 years of age.
3. All patients must have histologically confirmed adenocarcinoma of the rectum with pathologic material reviewed by the Department of Pathology at MDACC. The clinical stage must be T3, T4, or recurrent based on CT, MRI or EUS criteria.
4. All patients must have no distant metastatic disease on abdominopelvic CT scan performed with IV contrast. If the CT was performed outside of MDACC, the slice thickness is 7.5 mm. Criteria for pathologic enlargement of lymph nodes is > 15 mm on short axis dimension. If CT findings of lung, liver, or peritoneal metastases are equivocal, patients are eligible to participate.
5. The rectal tumor must be either palpable on digital rectal exam or the inferior edge of the tumor must be within 12 cm of the anal verge based on rigid proctoscopy.
6. Patients must have WBC > 4000 cells/mm3, ANC of >1500/L, platelets > 100,000/mm3, total serum bilirubin < 2.0 mg%, BUN < 30 mg%, creatinine < 1.5 mg% and/or creatinine clearance >30ml/min (estimated as calculated with Cockcroft-Gault equation). Note: In patients with moderate renal impairment (estimated creatinine clearance 30-50 mL/min) at baseline, a dose reduction to 75% of the capecitabine starting dose is recommended.
7. Hemoglobin of >9 gm/dL (may be transfused or receive Procrit to maintain or exceed this level)
8. Patients must have signed informed consent indicating that they are aware of the investigational nature of the study, and are aware that participation is voluntary.

Exclusion Criteria:

1. Known compromised renal or hepatic function.
2. Participation in any other experimental drug study.
3. AST or ALT >5 times upper limit of normal for subjects with documented liver metastases; >2.5 times the upper limit of normal for subjects without evidence of liver metastases.
4. Pregnant or lactating woman. Woman of childbearing potential with either a positive or no pregnancy test at baseline. Woman / men of childbearing potential not using a reliable contraceptive method. (Postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential). Patients must agree to continue contraception for 30 days from the date of the last study drug administration.
5. Any prior chemotherapy.
6. Any prior radiation therapy.
7. Serious, uncontrolled, concurrent infection(s) requiring IV antibiotics.
8. Treatment for other carcinomas within the last five years, except cure non-melanoma skin cancer and treated in-situ cervical cancer.
9. Clinically significant cardiac disease (e.g., uncontrolled hypertension [blood pressure of >160/110 mmHg on medication], any history of myocardial infarction, unstable angina), New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix H), unstable symptomatic arrhythmia requiring medication (subjects with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia are eligible), or grade II or greater peripheral vascular disease(see Appendix H).
10. Inability to to swallow oral medication.
11. Evidence of bleeding diathesis or coagulopathy, INR greater than or equal to 1.5.
12. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study; fine needle aspirations or core biopsies within 7 days prior to Day 0.
13. Proteinuria at baseline or clinically significant impairment of renal function Subjects unexpectedly discovered to have 1+ proteinuria at baseline should undergo a 24-hour urine collection, which must be an adequate collection and must demonstrate <500 mg of protein/24 hr to allow participation in the study (see appendix F).
14. Currently has serious, nonhealing wound, ulcer, or bone fracture.
15. Had aneurysms, strokes, transient ischemic attacks, and arteriovenous malformations within the past year.
16. Patients who have had an organ allograft.
17. Patients on Coumadin must be changed to Lovenox at least 1 week prior to starting capecitabine. Low dose (1 mg) Coumadin is allowed.
18. Patients taking Sorivudine or Brivudine A must be off of these drugs for 4 weeks. Patients taking cimetidine must have this drug discontinued. Ranitidine or a drug from another anti-ulcer class can be substituted for cimetidine if necessary. If patient is currently receiving allopurinol, must discuss with PI to see of another agent may substitute for it.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher H. Crane, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 4/21/05 through 8/31/07. All participants recruited at UT MD Anderson Cancer Center.
Groups:
- Avastin: Neoadjuvant therapy with radiotherapy (50.4 Gy in 28 fractions over 5.5 weeks), Avastin every 2 weeks (3 doses of 5 mg/kg), and capecitabine (900 mg/m2 orally twice daily only on days of radiation) followed by surgical resection.
Period: Overall Study
Arm/Group | Avastin
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Avastin
Number analyzed (Participants) | 25
Age Continuous [Mean (Full Range); unit: years] | 51 [34 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Local Tumor Response
Description: At follow-up evaluation after completion of neoadjuvant and surgical therapy, resected primary tumor classified based on routine pathology staining in the following manner: Pathologic Complete Response (no evidence of residual cancer); Microscopic Residual (no grossly detected disease, but evidence of microscopic residual disease); and Gross Residual Disease.
Time Frame: Baseline to approximately 5 Months (Following 28 days of treatment, chemotherapy and surgical resection of tumor)
Population: Intention to treat analysis method. Data examination conducted upon enrollment and evaluability of 25 patients.
Measure: Number; unit: Participants
Arm/Group | Avastin
Number analyzed (Participants) | 25
Participants
  Pathological Complete Response | 8
  Microscopic Residual (<10% viable tumor cells) | 6
  Gross Residual Disease | 11

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | Avastin
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 1/25
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avastin (N=25)
Amyloidosis (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No